CLINICAL TRIAL: NCT02564796
Title: Erythropoietin to Prevent Unnecessary Transfusions In Patients With Cyanotic Congenital Heart Disease - A Prospective Randomized Control Trial
Brief Title: Erythropoietin to Prevent Unnecessary Transfusions In Patients With Cyanotic CHD - A Prospective Control Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David Werho, MD, Assistant Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160871
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Cyanotic Congenital Heart Disease; Anemia; Cyanosis; Congenital Heart Disease
Keywords: Erythropoetin; Cyanotic Heart Disease; Transfusion; Congenital Heart Disease
MeSH Terms: conditions — Anemia; Cyanosis; Heart Defects, Congenital | interventions — Epoetin Alfa; Iron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Group II (non-treatment group): Patients in the treatment group will not receive any extra intervention outside of standard of care. They will receive iron supplementation for 6 weeks starting before 8 weeks of age, 1 week after their first procedure (surgery or heart catheterization). They will be followed for 14 weeks.
  Interventions: Drug: Iron
- Epoetin alfa and iron supplements (Experimental): Group I (treatment group): Patients in the treatment group will receive weekly EPO injections and iron supplementation for 6 weeks starting before 8 weeks of age, 1 week after their first procedure (surgery or heart catheterization) They will be followed for 14 weeks.
  Interventions: Drug: Epoetin Alfa and Iron

INTERVENTIONS:
Drug: Epoetin Alfa and Iron — Patients in the treatment group will receive weekly EPO injections and iron supplementation for 6 weeks starting before 8 weeks of age, 1 week after their first procedure (surgery or heart catheterization) They will be followed for 14 weeks.
  Other Names: No other name
  Arms: Epoetin alfa and iron supplements
Drug: Iron — Patients in the treatment group will not receive any extra intervention outside of standard of care. They will receive iron supplementation for 6 weeks starting before 8 weeks of age, 1 week after their first procedure (surgery or heart catheterization). They will be followed for 14 weeks.
  Other Names: No other name
  Arms: Control

SUMMARY:
Cyanotic congenital cardiac patients require higher hemoglobin concentrations (red blood cell levels) for optimal oxygen delivery to the body. Prophylactic erythropoietin (EPO) and iron can prevent and/or decrease the amount of blood transfusions needed in this population. We seek to investigate if EPO and iron make a clinically significant difference in the number of transfusions given to these patients and the morbidity associated with it.

DETAILED DESCRIPTION:
Congenital heart disease occurs in about 1% of all live births. Cyanotic cardiac lesions in particular are at risk for significant mortality and morbidity because of their reduced ability to provide adequate oxygenation to the body and the brain. Many experts believe that to have adequate oxygen carrying capacity that these infants should ideally have a hemoglobin level greater than 13 g/dL. Many of these patients require blood transfusions prior to surgery to provide adequate oxygenation. The cause for this is likely multifactorial including normal neonatal physiology, frequent lab draws, and co-morbidities. Although rare, the morbidity due to transfusions can be devastating to this population including transmitted infections, transfusion reactions, extra hospitalizations, and antigen sensitization that would complicate heart transplant if needed.

There are centers in the United States that have developed protocols using erythropoietin to minimize blood product transfusions before and after surgery, also referred to as "bloodless surgery". There have been retrospective studies evaluating the success of these protocols, but there are no randomized controlled prospective studies that the investigators have studying the effects of erythropoietin effects in patients with cyanotic heart disease in regards to transfusion prevention.

Congenital cyanotic cardiac patients require higher hemoglobin concentrations for optimal oxygen delivery. Prophylactic erythropoietin can prevent and/or decrease the amount of blood transfusions needed prior to surgery. The researchers seek to investigate if erythropoietin makes a clinically significant difference in the number of transfusions given to these patients and the morbidity associated with it.

ELIGIBILITY:
Inclusion Criteria

* Newborns less than 4 weeks old at diagnosis
* Gestational age >34 weeks
* Birth weight 2.2-4kg
* Cyanotic heart disease who have had a surgical shunt or a catheterization intervention that is equivalent to a shunt (patent ductus arteriosus stent, right ventricular outflow tract stent).
* Baseline hematocrit to be below <40%.
* Completes at least 1 injection in the study by 8 weeks of age.

Exclusion Criteria

* Infants diagnosed at greater than 4 weeks of age
* Gestation <34 weeks
* Birth weight <2.2 kg or >4kg
* Hematocrit >40%
* Newborns with acyanotic heart disease
* Infants with significant co-morbidities:

  * Renal failure (Creatinine > 2 standard deviations above age adjusted norm)
  * Hepatic failure (elevated AST/ALT levels > 2 standard deviations above age adjusted norm
  * Hemolytic disease
  * Hemoglobinopathies (Sickle-cell disease, Thalassemias)

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K Werho, MD, Principal Investigator — University of California, San Diego/Rady Children's Hospital San Diego
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donato H. Erythropoietin: an update on the therapeutic use in newborn infants and children. Expert Opin Pharmacother. 2005 May;6(5):723-34. doi: 10.1517/14656566.6.5.723. PMID 15934899
- [Background] Fearon JA, Weinthal J. The use of recombinant erythropoietin in the reduction of blood transfusion rates in craniosynostosis repair in infants and children. Plast Reconstr Surg. 2002 Jun;109(7):2190-6. doi: 10.1097/00006534-200206000-00002. PMID 12045535
- [Background] Maier RF, Obladen M, Muller-Hansen I, Kattner E, Merz U, Arlettaz R, Groneck P, Hammer H, Kossel H, Verellen G, Stock GJ, Lacaze-Masmonteil T, Claris O, Wagner M, Matis J, Gilberg F; European Multicenter Erythropoietin Beta Study Group. Early treatment with erythropoietin beta ameliorates anemia and reduces transfusion requirements in infants with birth weights below 1000 g. J Pediatr. 2002 Jul;141(1):8-15. doi: 10.1067/mpd.2002.124309. PMID 12091844
- [Background] Richard S, Brion JP, Couck AM, Flament-Durand J. Accumulation of smooth endoplasmic reticulum in Alzheimer's disease: new morphological evidence of axoplasmic flow disturbances. J Submicrosc Cytol Pathol. 1989 Jul;21(3):461-7. PMID 2477140

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 Patients who had been screened/consented for the study did not reach the minimum hematocrit threshold for enrollment and were therefore screen failures.
Period: Overall Study
Arm/Group | Control | Epoetin Alfa and Iron Supplements
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Epoetin Alfa and Iron Supplements | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Transfusions Needed
Description: Prophylactic erythropoietin can prevent and/or decrease the amount of blood transfusions needed prior to surgery. We seek to investigate if erythropoietin makes a clinically significant difference in the number of transfusions given to these patients and the morbidity associated with it during the period in which the subjects will be active in the study (from baseline to 14 weeks post initial injection). The primary aim will be assessed when all subjects have completed week 14 or discontinue early.
Time Frame: First 4 months of life
Population: The principal investigator discussed the study's future with the sub-investigators on the study and came to the conclusion to close the study due to low enrollment while also considering the financial costs to continue to run the study.
Arm/Group | Control | Epoetin Alfa and Iron Supplements
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Oxygen Saturation
Description: Often, cyanotic congenital heart defect neonates have prolonged initial hospital stays due to the inability to maintain acceptable oxygen saturations, and transition to adequate oral intake for appropriate weight gain. If the hospital stay is found to be shortened after starting erythropoietin, this may be of clinical and financial significance.
Time Frame: First 4 months of life
Population: as for outcome 1
Arm/Group | Control | Epoetin Alfa and Iron Supplements
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Hospitalizations
Description: The number of hospital readmissions (related to failure to thrive or cyanosis) may imply the overall clinical stability of a patient. Because these infants are at high risk for mortality at home, there are multiple reasons why they may be admitted to the hospital including clinically significant anemia which requires blood transfusions, poor weight gain, difficulty feeding, inadequate oxygen saturations, and illnesses. Each admission is stressful to the patient and their families. Having a normal hemoglobin level may have a role in preventing several of these factors, especially regarding failure to thrive or cyanosis.
Time Frame: First 4 months of life
Population: as for outcome 1
Arm/Group | Control | Epoetin Alfa and Iron Supplements
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Weight Gain
Description: The secondary outcome of weight gain is appropriate in the setting of infants as this variable has been used to monitor the ability to thrive and meet the body's metabolic demands. It is well established in pediatrics that the neonate and infant should gain 15-30 grams per day for optimal growth. Infants who are cyanotic already have a deficiency in meeting their metabolic demands due to a reduced oxygen carrying capacity. This is further complicated in the instance of anemia. Thus, infants may have an increased ability to optimize weight gain in the setting of normal, stable hemoglobin levels which may be achieved with erythropoietin.
Time Frame: First 4 months of life
Population: as for outcome 1
Arm/Group | Control | Epoetin Alfa and Iron Supplements
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Initial Discharge
Description: If the hospital stay is found to be shortened after starting erythropoietin, this may be of clinical and financial significance.
Time Frame: First 4 months of life
Population: as for outcome 1
Arm/Group | Control | Epoetin Alfa and Iron Supplements
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control | Epoetin Alfa and Iron Supplements
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The principal investigator discussed the study's future with the sub-investigators on the study and came to the conclusion to terminate the study early due to low enrollment while also considering the financial costs to continue to run the study. It would be highly improbable to be able to enroll 54 more patients with the amount of funding left in the grant. No subjects were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT02564796/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT02564796/ICF_001.pdf